CLINICAL TRIAL: NCT03548311
Title: Japanese Early-stage Clinical Trial of Ultra-high Dose Methylcobalamin for Amyotrophic Lateral Sclerosis: a Pivotal Phase 3 Randomized Controlled Study
Brief Title: Clinical Trial of Ultra-high Dose Methylcobalamin for ALS
Acronym: JETALS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Collaborators: University of Tokushima (Other)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 763
Record Dates: First submitted 2018-05-14; First posted 2018-06-07 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-02

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; motor neuron disease; Lou Gehrig's disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease | interventions — mecobalamin; Saline Solution

STUDY DESIGN:
Intervention Model Description: double-blinded randomized controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment Phase: Placebo (Placebo Comparator): intramuscular injection of saline solution
  Interventions: Drug: saline solution
- Treatment Phase: methylcobalamin (Active Comparator): intramuscular injection of methylcobalamin
  Interventions: Drug: methylcobalamin
- OLE Phase: methylcobalamin (Experimental): intramuscular injection of methylcobalamin
  Interventions: Drug: methylcobalamin
- Tsunagi Phase: methylcobalamin (Experimental): intramuscular injection of methylcobalamin
  Interventions: Drug: methylcobalamin

INTERVENTIONS:
Drug: methylcobalamin — Patients receive methylcobalamin 50mg intramuscular injection twice a week.
  Arms: OLE Phase: methylcobalamin; Treatment Phase: methylcobalamin; Tsunagi Phase: methylcobalamin
Drug: saline solution — Patients receive saline solution intramuscular injection twice a week.
  Arms: Treatment Phase: Placebo

SUMMARY:
To examine the clinical efficacy and safety of ultra-high dose (50mg, im, twice a week) methylcobalamin in retarding the progression of symptoms in amyotrophic lateral sclerosis (ALS) patients, we enroll ALS patients diagnosed by Updated Awaji Criteria within 12 months after the clinical onset. First they are followed for 12 weeks with Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) scores, and only those who exhibit drops of 1-2 points are allowed to enter into the test period. A total of 128 patients are randomized and the half having placebo. They are blindly evaluated for drops of ALSFRS-R in 16 weeks, as the primary outcome. After this, all subjects receive methylcobalamin.

ELIGIBILITY:
Inclusion Criteria:

Treatment and OLE Phase:

* ALS patients within 12 months after clinical onset at the entry
* Diagnosed based on updated Awaji criteria: definite, probably or laboratory supported probable
* Decline of ALSFRSR being 1 or 2 during observation period of 12 weeks
* Japanese Clinical Severity Scale 1 or 2
* Those who can visit the participating medical centers

Tsunagi Phase:

- The subjects for the Tsunagi phase are patients with ALS who are continuing the administration of this drug at the time of approval, and have obtained consent for the transition to the Tsunagi phase.

Exclusion Criteria:

Treatment and OLE Phase:

* Those who have tracheostomy
* Those who had NIPPV
* %FVC<60%
* Those who have Chronic Obstructive Pulmonary Disease (COPD)
* Those who have symptoms and signs of B12 deficiency
* Those who had edaravone less than 4 weeks prior to entry
* Those who changed the schedule and dosing of riluzole
* Those who have dementia
* Those who have the possibility of pregnancy
* Those who have serious respiratory or cardiac diseases
* Those who have malignancies
* Those who participated other clinical trials within 12 weeks
* Those who have allergies to B12 and related compounds

Tsunagi Phase:

Not applicable.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
Treatment Phase: ALSFRS-R | during 16 weeks of test period
  Drop of Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (maximum or normal 48 and minimum 0; higher values represent better condition)

SECONDARY OUTCOMES:
Treatment Phase: time to event | during 16 weeks of test period
  time from the randomization to the onset of any of the event (24-hour use of noninvasive respiratory support, use of invasive respiratory support, or death)
Treatment Phase: %Functional Vital Capacity (FVC) | during 16 weeks of test period
  changes of per cent Functional Vital Capacity
Treatment Phase: homocystein | during 16 weeks of test period
  changes of serum levels of homocystein
Treatment Phase: Manual Muscle Testing (MMT) | during 16 weeks of test period
  changes of sum of Medical Research Council scales of manual muscle testing, ranging 5 (normal), 4, 4+, 3, 2, 1, 0 (minimal) ( for analysis each is converted to 6, 5, 4, 3, 2, 1, 0) of the 11 muscles in the limbs (5x2) and neck(1)
Treatment Phase: Norris scale | during 16 weeks of test period
  changes of Norris scale (39 normal - 0 worst)
Treatment Phase: Grip Power | during 16 weeks of test period
  changes of sum of grip power in kilograms on both sides
Treatment Phase: 40-item Amyotrophic Lateral Sclerosis Assessment Questionnaire (ALSAQ-40) | during 16 weeks of test period
  changes of sum of ALSAQ-40 (40-item Amyotrophic Lateral Sclerosis Assessment Questionnaire) score (40 normal - 200 worst)

OTHER OUTCOMES:
Treatment Phase: safety | during 16 weeks of test period
  any adverse events during the treatment period
OLE Phase: time to event | up to 6 years 11 months
  time from the randomization to the onset of any of the event (24-hour use of noninvasive respiratory support, use of invasive respiratory support, or death)
OLE Phase: ALSFRS-R | up to 6 years 11 months
  Drop of ALSFRS-R Scale-Revised (maximum or normal 48 and minimum 0; higher values represent better condition)
OLE Phase: safety | up to 6 years 11 months
  any adverse events during the OLE period including laboratory tests and vital signs assessment.
Tsunagi Phase: time to event | up to 6 months
  time period from drug assignment to any of the event (24-hour use of noninvasive respiratory support, use of invasive respiratory support, or death)
Tsunagi Phase: ALSFRS-R | up to 6 months
  Drop of ALSFRS-R Scale-Revised (maximum or normal 48 and minimum 0; higher values represent better condition)
Tsunagi Phase: safety | up to 6 months
  any adverse events during the Tsunagi phase including laboratory tests and vital signs assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Ryuji Kaji, MD, Study Director — Tokushima University Hospital
Locations (16):
- Japan (16):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Miyoshi Neurological Clinic, Miyoshi, Hiroshima
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Kobe Central Munincipal Medical center, Kobe, Hyōgo
  - Ioh National Hospital, Kanazawa, Ishikawa-ken
  - Kitasato University East Hospital, Sagamihara, Kanagawa
  - Shiga Medical University Hospital, Ōtsu, Shiga
  - Chiba University Hospital, Chiba
  - Murakami Karindo Hospital, Fukuoka
  - Okayama University Hospital, Okayama
  - Tokushima University Hospital, Tokushima
  - Juntendo University Hospital, Tokyo
  - Toho University Hospital, Tokyo
  - Teikyo University Hospital, Tokyo
  - Tokyo Metropolitan Neurological Hospital, Tokyo
  - Wakayama Medical University Hospital, Wakayama

IPD SHARING:
Plan to Share IPD: Yes
anonymous data are available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: from October 1, 2017 till March 31, 2020
Access Criteria: those who have approval from Institutional Review Board (IRB)
URL: http://als-mecobalamin.org

REFERENCES:
- [Result] Ikeda K, Iwasaki Y, Kaji R. Neuroprotective effect of ultra-high dose methylcobalamin in wobbler mouse model of amyotrophic lateral sclerosis. J Neurol Sci. 2015 Jul 15;354(1-2):70-4. doi: 10.1016/j.jns.2015.04.052. Epub 2015 May 8. PMID 25982504
- [Result] Kaji R, Kodama M, Imamura A, Hashida T, Kohara N, Ishizu M, Inui K, Kimura J. Effect of ultrahigh-dose methylcobalamin on compound muscle action potentials in amyotrophic lateral sclerosis: a double-blind controlled study. Muscle Nerve. 1998 Dec;21(12):1775-8. doi: 10.1002/(sici)1097-4598(199812)21:123.0.co;2-v. PMID 9843082
- [Derived] Oki R, Izumi Y, Fujita K, Miyamoto R, Nodera H, Sato Y, Sakaguchi S, Nokihara H, Kanai K, Tsunemi T, Hattori N, Hatanaka Y, Sonoo M, Atsuta N, Sobue G, Shimizu T, Shibuya K, Ikeda K, Kano O, Nishinaka K, Kojima Y, Oda M, Komai K, Kikuchi H, Kohara N, Urushitani M, Nakayama Y, Ito H, Nagai M, Nishiyama K, Kuzume D, Shimohama S, Shimohata T, Abe K, Ishihara T, Onodera O, Isose S, Araki N, Morita M, Noda K, Toda T, Maruyama H, Furuya H, Teramukai S, Kagimura T, Noma K, Yanagawa H, Kuwabara S, Kaji R; Japan Early-Stage Trial of Ultrahigh-Dose Methylcobalamin for ALS (JETALS) Collaborators. Efficacy and Safety of Ultrahigh-Dose Methylcobalamin in Early-Stage Amyotrophic Lateral Sclerosis: A Randomized Clinical Trial. JAMA Neurol. 2022 Jun 1;79(6):575-583. doi: 10.1001/jamaneurol.2022.0901. PMID 35532908
- [Derived] Oki R, Izumi Y, Nodera H, Sato Y, Nokihara H, Kanai K, Sonoo M, Urushitani M, Nishinaka K, Atsuta N, Kohara N, Shimizu T, Kikuchi H, Oda M, Ikeda K, Nagai M, Komai K, Kojima Y, Kuzume D, Isose S, Shimohama S, Abe K, Ito H, Noda K, Ishihara T, Morita M, Shimohata T, Teramukai S, Kagimura T, Noma K, Yanagawa H, Kuwabara S, Kaji R; JETALS. The Japanese Early-Stage Trial of High-Dose Methylcobalamin for Amyotrophic Lateral Sclerosis (JETALS): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2018 Dec 21;7(12):e12046. doi: 10.2196/12046. PMID 30578206